CLINICAL TRIAL: NCT06126510
Title: A Single-arm, Multicenter, Open-label Phase IIa Clinical Study to Evaluate the Efficacy and Safety of VG161 in the Treatment of Advanced Bone and Soft Tissue Sarcoma
Brief Title: Clinical Study of VG161 in the Treatment of Advanced Bone and Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C206
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Single Arm (Experimental): VG161:1.0 × 10 ^ 8 PFU daily for 3 consecutive days on Days 1-3 of each cycle (D1-D3)
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell) — VG161:1.0×10^8PFU/day, intratumoral injection administration for 3 consecutive days, 28 days as a cycle
  Other Names: VG161

SUMMARY:
This study plans to use 1.0×108PFU/day per cycle, intratumoral injection administration for 3 consecutive days, and 28 days as a cycle. Tumor imaging evaluation was performed every 8±1 weeks from the first dose of C1D1 until an event that met the criteria for treatment discontinuation occurred.

DETAILED DESCRIPTION:
This study plans to use 1.0×108PFU/day per cycle, intratumoral injection administration for 3 consecutive days, and 28 days as a cycle. Tumor imaging evaluation was performed every 8±1 weeks from the first dose of C1D1 until an event that met the criteria for treatment discontinuation occurred. If the subject VG161 injection target lesion shrinks after treatment and can no longer receive intratumoral injection administration of this administered dose of VG161, after evaluation by the investigator, it is allowed to reduce the dosing dose or suspend the administration as appropriate according to the size of the injectable lesion. After the end of treatment, there will also be an end-of-treatment visit and a post-treatment safety visit. Subjects who end the study for reasons not attributable to disease progression will undergo imaging evaluation at the end of treatment (if no imaging evaluation is performed within 4 weeks) and have imaging every 3 months after the end of treatment until disease progression or death or initiation of new anti-tumor therapy (whichever occurs first) to assess the time to disease progression. After the end of treatment, the subjects will also receive survival follow-up once every 3 months, and the survival status of the subjects and subsequent anti-tumor therapy will be collected and recorded until death, loss to follow-up or 1 year after the last dose (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give informed consent to this study before the trial and voluntarily sign a written informed consent form.
* Age 18 to 75 years old (inclusive), gender is not limited.
* Patients with advanced bone and soft tissue sarcoma confirmed by histopathological or cytology, who are unresectable by surgery and have failed at least one standard treatment (among them, patients with Ewing sarcoma need to be patients without standard treatment).
* According to RECIST 1.1, it is determined that at least one CT examination shows measurable and meets the volume requirement for the first injection, superficial lesions are preferred, and tumor lesions that can be injected under ultrasound guidance can also be selected (the injected lesions are preferably major tumor burden lesions), and the longest diameter of the injected lesion at baseline (short diameter for lymph node lesions) > 1.5cm.
* Those who have a positive HSV-1 IgG or HSV-1 IgM antibody test result (HSV-1 IgM).
* ECOG physical status score of 0-1.
* Estimated survival time of more than 3 months.
* Have adequate organ function:

  1. Blood routine (no blood transfusion or colony-stimulating factor therapy within 14 days): ANC≥1.5×109/L, PLT≥75×109/L, Hb≥85g/L, lymphocyte count≥1.5×109/L (for lymphocyte count 0.8×109/L to 1.5×109/L at the discretion of the investigator);
  2. Liver function: TBIL ≤1.5×ULN, ALT≤3×ULN, AST≤3×ULN (ALT≤5×ULN and AST≤5×ULN are acceptable for patients with liver metastases);
  3. Renal function: Cr≤1.5×ULN, and creatinine clearance ≥45ml/min (calculated according to Cockcroft-Gault formula);
  4. Coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5×ULN, international normalized ratio (INR) ≤1.5×ULN.
* Eligible subjects (males and females) of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) for the duration of the trial and for at least 3 months after the last dose; Female patients of childbearing potential must have a negative blood pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor drugs within 4 weeks before the first use of study drugs, among which oral fluorouracils and small molecule targeted drugs are the first use of study drugs. Within the first 2 weeks or the 5 half-lives of the drug (whichever is longer).
* Have received other unmarketed clinical trial treatments within 4 weeks before using the study drug for the first time.
* Have undergone major organ surgery (excluding puncture biopsy) or experienced significant trauma within 4 weeks before taking the study drug for the first time.
* Patients who have received systemic corticosteroids (prednisone >10 mg/day or equivalent doses of similar drugs) or other immunosuppressants within 14 days before the first use of study drugs; Exceptions are the following: treatment with topical, ocular, intraarticular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids (≤10 mg prednisone equivalent) for prophylactic treatment (e.g., prevention of contrast media allergy).
* Have received vaccination within 4 weeks before the first use of study drugs.
* The adverse reactions of previous anti-tumor treatments have not returned to CTCAE 5.0 grade ≤1 (except for toxicities such as hair loss that the researcher has judged to have no safety risks).
* Patients with central nervous system metastasis or meningeal metastasis are not suitable for inclusion according to the investigator's judgment.
* With spinal cord compression, the researcher determines that the patient is not suitable for enrollment.
* In the period of recurrent infection of herpes simplex virus, with corresponding clinical manifestations, such as cold sores, herpetic keratitis, herpetic dermatitis, genital herpes, etc.
* Other uncontrolled active infections.
* Have a history of immunodeficiency, including positive HIV antibody test and Treponema pallidum antibody test.
* Patients with active chronic hepatitis B or active hepatitis C (except hepatitis B virus carriers, stable hepatitis B after drug treatment [negative HBV-DNA test or <50IU/ml] and cured hepatitis C patients [HCV RNA Tested negative]).
* Have a history of severe cardiovascular disease:

  1. Ventricular arrhythmias requiring clinical intervention;
  2. QTc interval>480ms;
  3. Acute coronary syndrome, congestive heart failure, stroke or other grade III or above cardiovascular events within 6 months before using the study drug for the first time;
  4. New York Heart Association (NYHA) cardiac function class ≥ class II or left ventricular ejection fraction (LVEF) <40%;
  5. Uncontrolled hypertension (systolic blood pressure ≥140mmHg, or diastolic blood pressure ≥90mmHg after treatment).
* Patients with active or past autoimmune diseases that may relapse (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (including but not limited to these diseases or syndromes, etc.); but does not include patients with clinically stable autoimmune thyroiditis, autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone; Type I diabetes on insulin; patients with vitiligo or childhood asthma/allergies that have resolved and do not require any intervention in adulthood.
* Have received immunotherapy and experienced immune-related adverse events (irAEs) such as immune-related pneumonia, myocarditis, etc., which may affect the safety of the trial medication as judged by the researcher.
* Known dependence on alcohol or drugs.
* People with mental disorders or poor compliance.
* Pregnant or lactating women.
* Patients with obvious symptoms and unstable pleural effusion, peritoneal effusion or pericardial effusion (those with stable clinical symptoms after treatment of pleural effusion, ascites or pericardial effusion can be included).
* The researcher believes that the subject has other serious systemic diseases or other reasons and is not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
ORR | through the study completion, an average of 2 year
  Objective response rate (ORR)
4-month PFS rate | through the study completion, an average of 2 year
  4-month Progression Free Survival (PFS) rate
6-month PFS rate | through the study completion, an average of 2 year
  6-month Progression Free Survival (PFS) rate

SECONDARY OUTCOMES:
DCR | through the study completion, an average of 2 year
  disease control rate (DCR)
PFS | through the study completion, an average of 2 year
  Progression Free Survival (PFS)
OS | through the study completion, an average of 2 year
  Overall Survival (OS)
DOR | through the study completion, an average of 2 year
  Duration of Response (DOR)
Immunological indicators | through the study completion, an average of 2 year
  Immunological parameters: peripheral blood lymphocyte subsets (CD3 +, CD4 +, CD8 +, CD4 +/CD8 + ratio, CD19 +, CD16 + CD56 + (NK) cells), cytokines (IL-12, IL-15, IL-6, TNF-α, IFN-γ);
6-month OS rate | through the study completion, an average of 2 year
  6-month Overall Survival (OS) rate
12-month OS rate | through the study completion, an average of 2 year
  12-month Overall Survival (OS) rate

CONTACTS AND LOCATIONS:
Overall Officials: Lu Xie, Medical PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No